CLINICAL TRIAL: NCT05878587
Title: Effects of Burger Allen Exercises on Pain, Range of Motion, and Disability in Knee Osteoarthritis With Type II Diabetes
Brief Title: Burger Allen Exercises in Knee OA With Type II Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/23/0109/Ayesha iftikhar
Record Dates: First submitted 2023-04-18; First posted 2023-05-26 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Knee Osteoarthritis; Type II Diabetes
Keywords: Buerger Allen exercises; Diabetes mellitus; Knee osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): thermotherapy+ TENS+ low intensity high repetition exercises and Buerger Allen.
  Interventions: Other: thermotherapy+ TENS+ low intensity high repetition exercises and Buerger Allen
- Group B control group (Active Comparator): Thermotherapy+ TENS+ low intensity high repetition exercises.
  Interventions: Other: thermotherapy+ TENS+ low intensity high repetition exercises

INTERVENTIONS:
Other: thermotherapy+ TENS+ low intensity high repetition exercises and Buerger Allen — Patient will be asked to lie down flat on the plinth with legs elevated from 45 degrees until the skin turns pale, it will take approximately 2 minutes to occur. Then the patient turns to sit at the edge of the plinth with feet hanging and doing the following exercises; dorsiflexion, plantar flexion, inversion, eversion, and flexion the extension of toes, this phase may also be maintained for 2 minutes. Finally, the patient lies flat with his leg rested in a horizontal position and covered with a warm blanket for about 5 minutes
  Arms: Group A
Other: thermotherapy+ TENS+ low intensity high repetition exercises — The intervention will be repeated 3 times per day and the posttest will be conducted 5th day using KOOS, NPRS and goniometer.
  Arms: Group B control group

SUMMARY:
There is a potential link between diabetes mellitus (DM) and severity of osteoarthritis .Type 2 diabetes is a part of the metabolic syndrome (Mets) accompanied by ageing and mechanical stress are also a risk factor to osteoarthritis. Every anatomical component of the joint demonstrated faster joint deterioration and elevated inflammation at microcellular environment of individuals with DM. Normal chondrocytes capacity to adapt to the local glucose level is impaired by OA and there is a significant risk of glucose toxicity and increased glucose absorption. The most dependable and effective treatment for mild to early joint osteoarthritis is exercise. Active free exercises i.e. Buerger Allen exercises are used as a conservative perfusion therapy because they rely on how gravity affects the smooth muscles in the valves. Synovial fluid supports the joint's ability to recover while also reducing inflammation and enhancing overall joint function. The aim of the study is to determine the effect of Buerger Allen exercise and low intensity high repetition exercises on pain, range of motion and disability in knee osteoarthritis with type 2 diabetes. The study would be randomized controlled trial. Total thirty-six subjects will be assigned randomly by using lottery randomization into two groups. Group A will receive conventional therapy and an additional Buerger Allen exercise while Group B will be a control group receiving only baseline treatment. Numeric pain rating scale (NPRS), Ankle Brachial Index, KOOS and Goniometer will be used as outcome measure tools for pain, range of motion and disability. Measure will be taken at baseline and at the end of treatment session. The collected data will be analyzed in Statistical Package for the Social Sciences (SPSS) 25.0.If data will be normally distributed then parametric if not normally distributed than non-parametric

DETAILED DESCRIPTION:
One of the most common joint conditions, osteoarthritis (OA), causes diarthrodial articular cartilage to deteriorate, which in turn causes disability in adults. Osteoarthritis (OA) and Type 2 diabetes mellitus (T2DM) are common illnesses whose prevalence is projected to increase. The association between diabetes mellitus and OA was originally identified in 1961.After adjusting for body mass index, type 2 diabetes was recently discovered to be an independent risk factor of severe OA, with a Hazard Ratio (HR) of 2.1. One of the most popular forms of exercise for diabetic patients is the Buerger Allen exercise, which improves lower extremity perfusion and alleviates symptoms in those with lower limbs arterial insufficiency by using postural changes, stimulation of peripheral circulation, and application of muscle contraction. It has been found that nurses can prevent foot ulcers and lower limb amputations by educating the public, screening high-risk individuals, and giving medical care.

ELIGIBILITY:
Inclusion Criteria:

* Both Genders from Age:45-65 year

Exclusion Criteria:

* Joint Instability

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-03-31 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
KOOS | 10 months
  An instrument to assess the patient's opinion about their knee and associated problems.
Numeric Pain Rating Scale | 10 months
  NPRS is based on 11-point numerical rating scale for determining pain intensity, 0(no pain) to 10(worst pain imaginable) pain intensity.

SECONDARY OUTCOMES:
Ankle Brachial Index | 10 months
  Ankle Brachial Index Will be measured with bp apparatus to measure Perfusion.

OTHER OUTCOMES:
Goniometer | 10 months
  A universal goniometer is an instrument that measures the available range of motion at a joint. Knee flexion and extension will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad sanaullah, Principal Investigator — Riphah International University
Locations (1):
- Tehsil headquarter hospital, Barnala, Azad Kashmir, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] WAINE H, NEVINNY D, ROSENTHAL J, JOFFE IB. Association of osteoarthritis and diabetes mellitus. Tufts Folia Med. 1961 Jan-Mar;7:13-9. No abstract available. PMID 13782559
- [Background] Schett G, Kleyer A, Perricone C, Sahinbegovic E, Iagnocco A, Zwerina J, Lorenzini R, Aschenbrenner F, Berenbaum F, D'Agostino MA, Willeit J, Kiechl S. Diabetes is an independent predictor for severe osteoarthritis: results from a longitudinal cohort study. Diabetes Care. 2013 Feb;36(2):403-9. doi: 10.2337/dc12-0924. Epub 2012 Sep 21. PMID 23002084
- [Background] Saw MM, Kruger-Jakins T, Edries N, Parker R. Significant improvements in pain after a six-week physiotherapist-led exercise and education intervention, in patients with osteoarthritis awaiting arthroplasty, in South Africa: a randomised controlled trial. BMC Musculoskelet Disord. 2016 May 27;17:236. doi: 10.1186/s12891-016-1088-6. PMID 27233479
- [Background] Mobasheri A, Neama G, Bell S, Richardson S, Carter SD. Human articular chondrocytes express three facilitative glucose transporter isoforms: GLUT1, GLUT3 and GLUT9. Cell Biol Int. 2002;26(3):297-300. doi: 10.1006/cbir.2001.0850. PMID 11991658
- [Background] Griffin TM, Huffman KM. Editorial: Insulin Resistance: Releasing the Brakes on Synovial Inflammation and Osteoarthritis? Arthritis Rheumatol. 2016 Jun;68(6):1330-3. doi: 10.1002/art.39586. No abstract available. PMID 26749517
- [Background] Rosa SC, Goncalves J, Judas F, Mobasheri A, Lopes C, Mendes AF. Impaired glucose transporter-1 degradation and increased glucose transport and oxidative stress in response to high glucose in chondrocytes from osteoarthritic versus normal human cartilage. Arthritis Res Ther. 2009;11(3):R80. doi: 10.1186/ar2713. Epub 2009 Jun 2. PMID 19490621
- [Background] Tsai TL, Manner PA, Li WJ. Regulation of mesenchymal stem cell chondrogenesis by glucose through protein kinase C/transforming growth factor signaling. Osteoarthritis Cartilage. 2013 Feb;21(2):368-76. doi: 10.1016/j.joca.2012.11.001. Epub 2012 Nov 11. PMID 23151458
- [Background] Aguiari P, Leo S, Zavan B, Vindigni V, Rimessi A, Bianchi K, Franzin C, Cortivo R, Rossato M, Vettor R, Abatangelo G, Pozzan T, Pinton P, Rizzuto R. High glucose induces adipogenic differentiation of muscle-derived stem cells. Proc Natl Acad Sci U S A. 2008 Jan 29;105(4):1226-31. doi: 10.1073/pnas.0711402105. Epub 2008 Jan 22. PMID 18212116
- [Background] Cramer C, Freisinger E, Jones RK, Slakey DP, Dupin CL, Newsome ER, Alt EU, Izadpanah R. Persistent high glucose concentrations alter the regenerative potential of mesenchymal stem cells. Stem Cells Dev. 2010 Dec;19(12):1875-84. doi: 10.1089/scd.2010.0009. Epub 2010 Sep 11. PMID 20380516
- [Result] Zaharia OP, Pesta DH, Bobrov P, Kupriyanova Y, Herder C, Karusheva Y, Bodis K, Bonhof GJ, Knitza J, Simon D, Kleyer A, Hwang JH, Mussig K, Ziegler D, Burkart V, Schett G, Roden M, Szendroedi J. Reduced Muscle Strength Is Associated With Insulin Resistance in Type 2 Diabetes Patients With Osteoarthritis. J Clin Endocrinol Metab. 2021 Mar 25;106(4):1062-1073. doi: 10.1210/clinem/dgaa912. PMID 33382877